CLINICAL TRIAL: NCT03311581
Title: The Feasibility of Propofol TCI in Hemodialysis Patients Undergoing Arteriovenous Shunt Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20170080
Record Dates: First submitted 2017-09-17; First posted 2017-10-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-05

CONDITIONS: End Stage Renal Disease; Hemodialysis Complication
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Propofol group (Experimental): propofol TCI plus brachial plexus block with ropivacaine 0.5% 30 to 40 ml
  Interventions: Drug: Propofol
- Sevoflurane group (Active Comparator): sevoflurane 2~4 % plus brachial plexus block with ropivacaine 0.5% 30 to 40 ml
  Interventions: Device: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol works by increasing GABA-mediated inhibitory tone in the CNS. Propofol decreases the rate of dissociation of the GABA from the receptor, thereby increasing the duration of the GABA-activated opening of the chloride channel with resulting hyperpolarization of cell membranes.
  Arms: Propofol group
Device: Sevoflurane — sevoflurane inhalation 2~4%
  Arms: Sevoflurane group

SUMMARY:
Written informed consent must be obtained before any study specific procedures are undertaken. Informed consent will be obtained during pre-operative assessment.

DETAILED DESCRIPTION:
The investigators will recruit 80 patients undergoing AV shunt surgery. All patients will receive general anesthesia and brachial plexus block. Patients will be randomly allocated into two groups. Study and control group received propofol target-controlled infusion (TCI) and inhaled anesthetics as anesthesia maintenance, respectively. Main outcomes will be assessed by perioperative blood pressure, heart rate, respiratory rate, end-tidal CO2, analgesics dosage, pain intensity and perioperative adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Uremic adult(over20-year-old)patients under going arteriovenous (AV) shunt surgery

Exclusion Criteria:

* one of below systemic diseases; chronic pulmonary, cardiac diseases(such as COPD, asthma, acute myoischemia), hepatic co-mobility(such as liver cirrhosis), morbid obesity, alcoholism, allergy to propofol and inhaled anesthetics, the women who are pregnant or breastfeeding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | The blood pressure change between baseline, post-induction 3mins, operation start, post-operation 10 mins,post-operation 30 mins,post-operation 1 hour,post-operation 2 hours, end of surgery, recovery room, up to 4 hours
  Systolic blood pressure, diastolic blood pressure

SECONDARY OUTCOMES:
analgesics dosage | The amount of analgesics dosage use at recovery room,an average of 4 hours
  post-operation analgesics dosage
Change in pain intensity | The pain intensity change at recovery room, post-operation day 1, post-operation day 2
  Visual Analog Score for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan